CLINICAL TRIAL: NCT00684736
Title: Tryptophan, Serotonin and Kynurenine in Septic Shock
Acronym: TSK
Status: Completed | Type: Observational
Sponsor: Versailles Hospital (Other)
Responsible Party: Henry-Lagarrigue Matthieu/MD, Intensive Care Unit
Other Study IDs: TSK Sepsis
Record Dates: First submitted 2008-05-22; First posted 2008-05-28 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2008-05

CONDITIONS: Shock, Septic
Keywords: septic shock; shock; serotonin; kynurenine; tryptophan
MeSH Terms: conditions — Shock, Septic; Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Septic shock is a major cause of mortality and morbidity worldwide. Serotonin (5-HT) is released by activated platelets into the circulation, and is mediator of endothelial dysfunction. 5-HT metabolism is known in immune system via specific 5-HT receptor, also in effects on the peripheral nervous system. Kinetic of 5-HT, tryptophan, kynurenine, MAO activity and IDO activity in human septic shock was never investigated.

ELIGIBILITY:
Inclusion Criteria:

* Age above or equal to 18 years
* Strong presumption clinical sepsis
* Need for mechanical ventilation
* Body temperature above 38°C or below 36°C
* Heart rate above 90 bpm
* Systolic blood pressure of <90mm Hg despite adequate fluid replacement or a need for vasopressors less than 3 hours
* Presence of at least one of the following criteria:

  * Ratio of arterial oxygen tension over inspired fraction of oxygen of less than 300 mm Hg
  * Urinary output below 0.5 mL per kg of bodyweight per h or below 30 mL/h (for at least 1 h)
  * Arterial lactate concentration above 2 mmol/L
* Consent signed

Exclusion Criteria:

* Age below 18 years
* Pregnancy
* Underlying disease with a poor prognosis, a life expectancy of less than 24 hours
* Depression or melancholy
* Neuropsychiatric diseases: Seizure, manic psychosis, Migraine, or Drug addiction
* Neuroendocrine tumors
* Obstructive cardiomyopathy or acute myocardial ischaemia
* Pulmonary embolism
* Advanced stage cancer, malignant haemopathy, or AIDS with a decision to withhold or withdraw aggressive therapies
* Inclusion in another clinical trial
* Patient who receive before inclusion one of the following treatment known to modify serotonin level: almotriptan, amitriptyline, amoxapine, citalopram, clomipramine, clozapine, desipramine, dihydroergotamine, dolasetron, dosulepin, doxepin, eletriptan, ergotamine, flunarizine, fluoxetine, fluvoxamine, granisetron, imipramine, indoramin, interferon Alfa, interferon alfacon-1, interferon beta, iproniazid, maprotiline, methysergide, mianserin, Milnacipran, mirtazapine, moclobemide, naratriptan, olanzapine, ondansetron, oxetorone, paroxetine, pizotifen, risperidone, sertraline, sumatriptan, tianeptine, trimipramine, tropisetron, venlafaxine,viloxazine, zolmitriptan.
* No consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were 18 years of age or older and had been hospitalized in our ICU were prospectively enrolled in the study if they met all eligibility criteria. Inclusion criteria were clinical evidence of infection, evidence of a systemic response to infection, and the onset of shock within the previous 3 hours.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2004-06; Primary Completion 2007-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Kinetics of 5-HT, 5-HIAA, kynurenine, tryptophan, HVA, VMA, DOPAC, Oestradiol, Cotinine and vasopressors | Day-1, Day-2, Day-3, Day-7 and Day-14

SECONDARY OUTCOMES:
Mortality | 28-day

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Bédos, MD, PhD, Study Chair — Versailles Hospital; Odile Spreux-Varoquaux, PhD, Study Director — Versailles Hospital; Matthieu Henry-Lagarrigue, MD, Principal Investigator — Versailles Hospital
Locations (1):
- CH Versailles - André Mignot Hospital, Le Chesnay, France

REFERENCES:
- [Derived] Troche G, Henry-Lagarrigue M, Soppelsa F, Legriel S, Yehia A, Bruneel F, Bedos JP, Spreux-Varoquaux O. Tryptophan pathway catabolites (serotonin, 5-hydroxyindolacetic acid, kynurenine) and enzymes (monoamine oxidase and indole amine 2,3 dioxygenase) in patients with septic shock: A prospective observational study versus healthy controls. Medicine (Baltimore). 2020 May;99(19):e19906. doi: 10.1097/MD.0000000000019906. PMID 32384433